CLINICAL TRIAL: NCT06794164
Title: Immediate Skin-To-Skin Care For Preterm Infants After Birth
Acronym: eSCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1309/2024
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Effect of Skin to Skin Care in Preterm Neonates; Skin to Skin Care
Keywords: skin to skin care; preterm neonates
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early skin-to-skin care (Experimental): Intervention group
  Interventions: Procedure: skin to skin care
- Standard care group (Active Comparator): Control group
  Interventions: Procedure: Standard Care (in control arm)

INTERVENTIONS:
Procedure: skin to skin care — skin to skin care of preterm infants with their parents immediately after birth
  Arms: Early skin-to-skin care
Procedure: Standard Care (in control arm) — skin to skin care within 24 hours after birth
  Arms: Standard care group

SUMMARY:
The standard procedure in our centre for preterm neonates is to enable skin-to-skin (SSC) contact within 24 hours after birth. As early SSC immediately after birth might provide numerous positive effects for mothers and their preterm neonates, the objective of this study is to evaluate the feasibility, the safety and the effect of skin-to-skin contact immediately after birth in preterm neonates born with gestational age between 26+0 and 32+0 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 26+0 and 32+0 weeks
* Written parental informed consent

Exclusion Criteria:

* No intention of full life support
* Severe congenital malformation

Ages: 0 Minutes to 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-02-03 (Estimated); Study Completion 2027-02-03 (Estimated)

PRIMARY OUTCOMES:
vital parameter: Heart rate | during the first 2 hours after birth
vital parameter: Oxygen saturation | during the first 2 hours after birth
  in percent
vital parameter: blood pressure | during the first 2 hours after birth
  systolic, diastolic and mean blood pressure
vital parameter: Temperature | during the first 2 hours after birth

SECONDARY OUTCOMES:
blood sugar | 1 hour after birth
  capillary blood sugar measured 1 hour after birth
FiO2 (Fraction of inspired oxygen) | during first 2 hours after birth
  Need of oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No
It is single center study